CLINICAL TRIAL: NCT05839626
Title: First-in-human, Open-label Phase 1/2 Study to Investigate Safety and Efficacy of SAR445514, an NKcell Engager (NKCE) Targeting B-cell Maturation Antigen (BCMA) in Monotherapy in Participants With Relapsed/Refractory Multiple Myeloma (RRMM) and in Relapsed/Refractory Light-chain Amyloidosis (RRLCA)
Brief Title: A Study to Investigate Safety and Efficacy With SAR445514 in Participants With Relapsed/Refractory Multiple Myeloma (RRMM) and Relapsed/Refractory Light-chain Amyloidosis (RRLCA)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Early discontinuation based on sponsor decision not driven by any safety concerns.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCD17710; U1111-1279-2985 (Registry Identifier: ICTRP); 2022-502057-33-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-03-31; First posted 2023-05-03 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Relapsed/Refractory Multiple Myeloma; Amyloid Light-chain Amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- SAR445514 RRMM Dose escalation phase (Part 1a) (Experimental): SAR445514 will be administered to participants with relapsed/refractory multiple myeloma (RRMM) using subcutaneous route (SC)
  Interventions: Drug: SAR445514
- SAR445514 RRLCA Dose escalation phase (part 1b) (Experimental): SAR445514 will be administered to participants with relapsed/refractory light chain amyloidosis (RRLCA)) using subcutaneous route (SC)
  Interventions: Drug: SAR445514
- SAR445514 Dose level A (part 2) (Experimental): SAR445514 will be administered to participants with relapsed/refractory multiple myeloma (RRMM) using subcutaneous route (SC)
  Interventions: Drug: SAR445514
- SAR445514 Dose level B (part 2) (Experimental): SAR445514 will be administered to participants with relapsed/refractory multiple myeloma (RRMM) using subcutaneous route (SC)
  Interventions: Drug: SAR445514
- SAR445514 RRMM Dose expansion (part 3a) (Experimental): SAR445514 will be administered to participants with relapsed/refractory multiple myeloma (RRMM) using subcutaneous route (SC)
  Interventions: Drug: SAR445514
- SAR445514 RRLCA Dose expansion (part 3b) (Experimental): SAR445514 will be administered to participants with relapsed/refractory light chain amyloidosis (RRLCA) using subcutaneous route (SC)
  Interventions: Drug: SAR445514

INTERVENTIONS:
Drug: SAR445514 — Powder for solution for injection. Sub Cutaneous administration.

SUMMARY:
This is a first-in-human (FIH) Phase 1/Phase 2 study for evaluating SAR445514 in monotherapy in participants with relapsed/refractory multiple myeloma (RRMM) and relapsed/refractory light chain amyloidosis (RRLCA).

The study will comprise 3 parts:

A dose escalation phase (Part 1) in RRMM participants (Part 1a) that will evaluate several doses administered to determine 2 doses that will be tested in the dose optimization part.

A dose escalation will also be done in RRLCA participants (Part 1b) but started sequentially after the end of the dose escalation in RRMM participants. This dose escalation will evaluate the 2 doses planned to be used in dose optimization in RRMM, to ensure those doses are safe also for RRLCA participants.

A dose optimization phase (Part 2) that will be evaluating 2 doses determined from Part 1 to determine the preliminary recommended Phase 2 dose (pRP2D) and schedule for SAR445514 in RRMM.

A dose expansion phase (Part 3) that will evaluate the preliminary efficacy of pRP2D and schedule for SAR445514 in RRMM (Part 3a) and RRLCA (Part 3b).

Approximately 111 participants will be enrolled and treated by study intervention and separated as such:

Part 1a: Approximately 30 to 40 participants Part 1b: Approximately 6 to 12 participants Part 2: Approximately 30 participants Part 3a: Approximately 15 participants Part 3b: Approximately 14 participants

DETAILED DESCRIPTION:
The duration of the study for a participant will include A screening period: up to 28 days prior day 1 of cycle 1 (C1D1) A treatment period: enrolled participants will receive administration of 4 weeks cycles of SAR445514 subcutaneously.

The End of treatment visit will occur 30 days (+/- 7 days) from last investigational medicinal product (IMP) administration or prior initiation of further therapy, whichever comes first.

The follow-up period will continue until death, participant's request to discontinue study, final Overall Survival analysis or upon cancellation of survival follow-up at the discretion of the Sponsor at any timepoint.

ELIGIBILITY:
Inclusion Criteria:

Participants must have a documented diagnosis of multiple myeloma (Part 1a, 2, and 3a) or light chain amyloidosis (Part 1b and 3b).

Participants with RRMM (Part 1, 2, and 3a)

* Participants with measurable disease for RRMM
* Participants with MM must have received at least 2 prior lines of therapy which must include at least 2 consecutive cycles of a second or third generation immunomodulator, steroid, proteasome inhibitor and anti-CD38 monoclonal antibody (MoAb).
* Participants must have documented evidence of progressive disease (PD), as per IMWG 2016 criteria.

Participants with RR LCA (Part 1b and 3b) must have received at least 1 prior line of treatment comprising at least 1 proteasome inhibitor.

* Participants with measurable disease according to ISA 2012.
* Participants must have documented evidence of progressive disease (PD), as per ISA 2012 criteria.
* One or more organ impacted by amyloidosis as per National comprehensive cancer network (NCCN) guidelines.

For dose escalation, body weight within 40 to 120 kg

Capable of giving signed informed consent

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical conditions

* Primary refractory MM defined as participants who never achieved at least a minimal response with any treatment during the disease course
* Second primary malignancy

Participants with RRMM (Part 1a, 2, and 3a)

* For MM participants, primary systemic LCA and plasma cell leukemia
* For MM participants, congestive heart failure (New York Heart Association [NYHA]) Grade ≥II; cardiomyopathy, active ischemia, or any other uncontrolled cardiac condition

Participants with RR LCA (Part 1b and 3b)

* For LCA participants, evidence of clinically significant cardiovascular condition, defined as one or more of the following:

  1. N-terminal prohormone of brain natriuretic peptide (NT-proBNP) >8500 ng/mL
  2. New York Heart Association (NYHA) classification III or IV heart failure
  3. Heart failure that, in the opinion of the Investigator, is not primarily related to LCA cardiomyopathy (including, but not limited to, ischemic heart disease, uncorrected valvular disease, infections)
  4. Prior event (history) in the last 6 months of acute coronary syndrome, myocardial infarction or unstable angina as well as participants who during the last 6 months experienced a percutaneous cardiac intervention with stent and/or a coronary artery bypass
  5. Hospitalization in the last 4 weeks prior to treatment related to a cardiovascular event
  6. Participants with prior history of arrhythmia and/or cardiac conduction disorders for which a pacemaker or an implantable cardioverter defibrillator (ICD) is required but has not been placed. This includes, but may not be limited to, sustained ventricular tachycardia, association of an atrioventricular, or sinoatrial nodal dysfunction
* For LCA participants, a systolic blood pressure <100 mmHg or a diastolic blood pressure <55 mmHg.
* For LCA participants: previous or current diagnosis of symptomatic MM, including the presence of lytic bone disease, plasmacytomas, ≥60% plasma cells in the BM, or hypercalcemia.

All participants

* Uncontrolled infection within 14 days prior to study treatment.
* Known acquired immunodeficiency syndrome-related illness or known human immunodeficiency virus (HIV) disease requiring antiviral treatment or active hepatitis A (defined as positive hepatitis A antigen or positive IgM); HIV serology at screening will be tested for participants in countries where it is required by local regulations.
* Uncontrolled or active hepatitis B virus (HBV) infection: participants with positive B surface antigen (HBsAg) and/or HBV deoxyribonucleic acid (DNA)
* Active hepatitis C virus (HCV) infection: positive HCV ribonucleic acid (RNA) and negative anti-HCV.

Prior/concomitant therapy

* Any anti-MM drug treatment within 14 days before study treatment
* Prior allogenic hematopoietic stem cell (HSC) transplant with active graft-versus-host disease (GvHD) (GvHD any grade and/or being under immunosuppressive treatment within the last 2 months prior to first IMP).
* Any major procedure within 14 days before the initiation of the study treatment
* Administration of an anti-CD38 monoclonal antibody (isatuximab or daratumumab) less than 90 days prior to the first administration of study treatment.
* Administration of an anti-BCMA agent (including, but not limited to, CAR T-cells, TCEs, antibody drug conjugate) less than 21 days prior to the administration of study treatment.
* Unresolved toxicities from prior anticancer therapy, defined as not having resolved to CTCAE Version 5.0 Grade 1, at the exception of residual Grade 2 peripheral neurotoxicity related to bortezomib and/or thalidomide and considered as stable.
* Participants with a contraindication to dexamethasone.

Prior/concurrent clinical study experience

* Received any other investigational drugs or prohibited therapy for this study within 28 days or 5 half-lives from study treatment, whichever is shorter

Diagnostic assessments

* Hemoglobin <8 g/dL (5.0 mmol/L)
* Platelets <50 × 10^9/L (not permissible to transfuse a participant within 1 week prior to the screening platelet count to reach this level).
* Absolute neutrophil count (ANC) <1000 μL (1 × 10^9/L).
* Creatinine clearance <30 mL/min (Modification of Diet in Renal Disease Formula).
* Total bilirubin >1.5 × upper limit of normal (ULN) (unless the subject has documented Gilbert syndrome in which case direct bilirubin should not be >2.5 × ULN).
* Aspartate aminotransferase (AST/SGOT) or Alanine aminotransferase (ALT/SGPT) >2.5 × ULN.
* Participants with Grade 3 or 4 hypercalcemia (corrected serum calcium of >12.5 mg/dL; >3.1 mmol/L; ionized calcium >1.6 mmol/L; or requiring hospitalization) will not be eligible unless participants recover to Grade 2 or less under anti-hypercalcemia treatment.

Other exclusions

* Individuals accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalized
* Participant not suitable for participation, whatever the reason, as judged by the Investigator
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Dose escalation (part 1a - RRMM) Presence of dose limiting toxicities (DLT) | Cycle 1 - 4 weeks per cycle
  DLTs will be defined using NCI CTCAE version 5.0 or ASTCT criteria for CRS or ICANS.
Dose escalation (part 1a - RRMM) Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | From Baseline to end of follow-up (approx. 15 months)
  Presence of TEAEs, SAEs, and lab abnormalities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading
Dose optimization (part 2 - RRMM) Overall response rate (ORR) | Cycles 1 to 4 - 4 weeks per cycle
  ORR is defined as the proportion of participants with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) according to the 2016 International Myeloma Working Group (IMWG) criteria, after the last participant is treated for at least 4 cycles or prematurely discontinued.
Dose escalation (part 1b - RRLCA) Presence of dose limiting toxicities (DLT) at cycle 1 | Cycle 1 - 4 weeks per cycle
Dose escalation (part 1b - RRLCA) Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | From baseline to end of follow-up (approx. 15 months)
Dose expansion (part 3 - RRMM) Overall response rate (ORR) | Cycles 1 to 4 - 4 weeks per cycle
  ORR is defined as the proportion of participants with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) according to the 2016 International Myeloma Working Group (IMWG) criteria.
Dose expansion (part 3-RRLCA) Hematological response (HR) | Cycles 1 to 4 - 4 weeks per cycle
  HR is defined as the proportion of participants with sCR, CR, VGPR, and PR according to the European society of hematology/International society of hematology working group guidelines.

SECONDARY OUTCOMES:
Dose escalation (part 1 - RRMM) Overall response rate (ORR) | Cycle 1 to first progressive disease or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  ORR defined as the proportion of participants with sCR, CR, VGPR, and PR according to the 2016 IMWG criteria.
Dose optimization (part 2 - RRMM) Presence of dose limiting toxicities (DLT) | Cycles 1 to 4 - 4 weeks per cycle
Dose optimization (part 2 - RRMM) Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | From first dose of study treatment up to 30 days after last dose of study treatment (approx. 1 year with cycle of 28 days)
  Treatment-emergent adverse events (AEs) are defined as AEs that develop, worsen, or become serious during the treatment period. The treatment period is defined as the time from first dose of study treatment up to 30 days after last dose of study treatment.
Dose optimization & expansion (Part 2 & Part 3a - RRMM) Very Good Partial Response (VGPR) or Better Rate | Cycle 1 to first progressive disease or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  VGPR is defined as the proportion of participants with sCR, CR, and VGPR according to the 2016 IMWG criteria.
Dose optimization & expansion (Part 2 & Part 3a - RRMM) Duration of response (DOR) | Cycle 1 to first progressive disease or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  DOR is defined as the time from the date of the first response to the date of the first occurrence of progressive disease (PD as determined by the investigator or death from any cause, whichever happens first. DOR is determined only for participants who have achieved a response (PR or better).
Dose optimization & expansion (Part 2 & Part 3a - RRMM) Time to first response (TT1R) | Cycle 1 to first progressive disease or end of treatment whichever comes first (approx. 1 year with cycle of 28 days)
  TT1R is defined as the time from the date of the first response to the date of the first occurrence of progressive disease (PD as determined by the investigator or death from any cause, whichever happens first. DOR is determined only for participants who have achieved a response (PR or better).
Dose optimization & expansion (Part 2 & Part 3a -RRMM) Time to best response (TTBR) | Cycle 1 to first progressive disease or end of treatment whichever comes first (approx. 1 year with cycle of 28 days)
  TTBR is defined as the time from the first administration of the IMP to the date of first occurrence of best overall response (PR or better that is subsequently confirmed.
Dose optimization & expansion (Part 2 & Part 3a - RRMM) Progression free survival (PFS) | Cycle 1 to first progressive disease or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  PFS is defined as the time from the date of the first administration of the IMP to the date of first documentation of progressive disease or the date of death from any cause, whichever comes first. Responses will be determined according to IMWG criteria. Progression based on paraprotein will be confirmed based on two consecutive assessments.
Dose optimization & expansion (Part 2 & Part 3a - RRMM) Overall survival (OS) | Cycle 1 to end of follow-up or death (approx. 15 months with cycle of 28 days)
  OS is defined as the time from the date of the first administration of the IMP to death from any cause
Dose optimization & expansion (Part 2 & Part 3a - RRMM) Clinical benefit rate (CBR) | Cycle 1 to first progressive disease or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  CBR is the rate of participants with confirmed CR or PR at any time or stable disease (SD) of at least 6 months from the first IMP administration determined by the Investigator per IMWG 2016 criteria.
Dose escalation (part 1b - RRLCA) Overall Hematological Response (OHR) | Cycle 1 to first progressive disease or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  OHR is defined as the proportion of participants with CR, VGPR, and PR according to the International Society of Amyloidosis guidelines (ISA 2012).
Dose extension (part 3b - RRLCA) Hematological complete response rate (HCR). | Cycle 1 to first progressive disease or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  HCR is defined as the proportion of participants with complete response according to the ISA 2012.
Dose extension (part 3b - RRLCA) Hematological very good partial response rate or better (HVGPR) | Cycle 1 to first progressive disease or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  HVGPR defined as proportion of participants with very good partial response and CR as per ISA 2012 criteria
Dose expansion (part 3b - RRLCA) Overall survival (OS) | Cycle 1 to death or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  OS is defined as the time from the date of study entry to death from any cause.
Dose expansion (part 3b - RRLCA) Progression-Free Survival (PFS) | Cycle 1 to first progressive disease (organ or hematological) or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  PFS is defined as time from the time from the first administration of the IMP to any of the following: hematological progression, major organ progression (cardiac, kidney or liver) according to ISA 2012 criteria or death by any cause.
Dose expansion (part 3b - RRLCA) Time to first hematological response (TT1HR) | Cycle 1 to first progressive disease or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  TT1HR is defined as the time from the first administration of the IMP to the date of first hematological response (PR or better) that is subsequently confirmed.
Dose expansion (part 3b - RRLCA) Duration of hematological response (DOHR) | Cycle 1 to first progressive disease or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  DOHR is defined as time from the time from the first administration of the IMP to any of the following: hematological progression, major organ progression (cardiac, kidney or liver) according to ISA 2012 criteria or death by any cause.
Dose expansion (Part 3 - RRMM & RRLCA) Percentage of participants experiencing treatment-emergent adverse events (TEAEs) | From first dose of study treatment up to 30 days after last dose of study treatment (approx. 15 months with cycle of 28 days)
  Treatment-emergent adverse events (AEs) are defined as AEs that develop, worsen, or become serious during the treatment-emergent period.
Incidence rate of infusion associated reactions (IARs) | From cycle 1 to end of treatment (approx. 1 year with cycle of 28 days)
Incidence rate of injection site reactions (ISR) | From cycle 1 to end of treatment (approx. 1 year with cycle of 28 days)
Incidence of laboratory abnormalities | From cycle 1 to end of follow-up (approx. 15 months with cycle of 28 days)
Assessment of pharmacokinetics (PK) parameter of SAR445514: Ctrough | From cycle 1 to end of treatment (approx. 1 year with cycle of 28 days)
Assessment of pharmacokinetics (PK) parameter of SAR445514: AUClast | From cycle 1 to end of treatment (approx. 1 year with cycle of 28 days)
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to time of the last concentration observed above the lower limit of quantification (ie, Clast)
Assessment of pharmacokinetics (PK) parameter of SAR445514: Cmax | From cycle 1 to end of treatment (approx. 1 year with cycle of 28 days)
  Maximum observed concentration
Assessment of pharmacokinetics (PK) parameter of SAR445514: Tmax | From cycle 1 to end of treatment (approx. 1 year with cycle of 28 days)
  First time to reach Cmax
Incidence of anti-drug antibody (ADA) against SAR445514 | From cycle 1 to end of treatment (approx. 1 year with cycle of 28 days)
Dose extension (Part 3 - RRMM & RRLCA) Minimum Residual Disease (MRD) negativity rate | Cycle 1 to first progressive disease or end of follow-up whichever comes first (approx. 15 months with cycle of 28 days)
  MRD status in participants with response of VGPR or better

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- Australia (2):
  - Investigational Site Number : 0360001, Wollongong, New South Wales
  - Investigational Site Number : 0360002, Richmond, Victoria
- Belgium (4):
  - Institut Jules Bordet_Site Number : 0560002, Anderlecht
  - Het Ziekenhuisnetwerk Antwerpen vzw - ZNA Middelheim_Site Number : 0560001-2, Antwerp
  - Het Ziekenhuisnetwerk Antwerpen vzw - ZNA Cadix_Site Number : 0560001-1, Antwerp
  - Investigational Site Number : 0560001, Antwerp
- Czechia (2):
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2030001, Ostrava
- Investigational Site Number : 3480001, Budapest, Hungary
- Investigational Site Number : 3800001, Rozzano, Lombardy, Italy
- Spain (3):
  - Hospital Universitario Marqués de Valdecilla_Site Number : 7240001, Santander, Cantabria
  - Institut Catala d´oncologia - Badalona_Site Number : 7240002, Badalona, Catalonia
  - HOSPITAL CLINIC i PROVINCIAL BARCELONA_Site Number : 7240003, Barcelona
- United Kingdom (3):
  - Investigational Site Number : 8260003, Birmingham
  - Investigational Site Number : 8260002, London
  - Investigational Site Number : 8260001, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.